CLINICAL TRIAL: NCT07192705
Title: An Observational Cross-sectional Study Exploring Differences in Health Between People With Non-Tuberculous Mycobacteria Pulmonary Disease and People With Bronchiectasis Without NTM Pulmonary Infection.
Brief Title: Health Impact of Non-Tuberculous Mycobacteria Pulmonary Disease (NTM-PD)
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 178013; IRAS (Other: 348528)
Record Dates: First submitted 2025-08-11; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Non-Tuberculous Mycobacteria Pulmonary Disease; Bronchiectasis
Keywords: Non-Tuberculous Mycobacteria Pulmonary Disease; NTM-PD; Non-Tuberculous Mycobacteria Lung Disease; Health Impact of NTM-PD; Bronchiectasis; NTM-LD; Bronchiectasis without NTM-PD; Non-Pharmacological Intervention
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Tuberculous Mycobacteria-Pulmonary Disease (NTM-PD): People diagnosed with NTM-PD
- Bronchiectasis: People diagnosed with bronchiectasis but no evidence for NTM pulmonary infection

SUMMARY:
Nontuberculous mycobacteria (NTM) are environmental organisms found in soil and water. The majority do not cause human disease. When they do, this is mostly as a chronic lung infection in people with long-term lung problems such as chronic obstructive pulmonary disease (COPD), bronchiectasis, or cystic fibrosis. The number of people with NTM pulmonary disease (PD) is increasing, and its management can be complex, requiring prolonged treatment with multiple, often toxic, drugs in someone who may already be frail.

Non-drug approaches, such as airway clearance techniques, structured exercise, nutritional support and psychological care are used to help manage bronchiectasis and COPD. However, there is limited evidence about their benefit in people with NTM-PD. Also, it is not clear whether these patients' health needs are different from people with bronchiectasis alone.

The investigators want to identify the most important symptoms encountered by people with NTM-PD and patient preferences for care. The study also aims to explore whether the need for non-drug measures differs between people with and without NTM-PD who have other underlying lung disease.

The research will take place at one NHS centre and involve a single assessment of 40 people with NTM-PD not using specific antibiotics to treat their NTM and 40 people with bronchiectasis but no evidence for NTM. Following consent, and mainly using questionnaires, participants will be asked about their physical and mental health, and nutritional status. Exercise capacity, muscle strength and body muscle/fat composition will also be assessed using simple tests. The total time required will be a maximum of one hour. Recruitment to the study will last around six months.

The results will help improve understanding of specific needs of people with NTM-PD and guide clinically relevant research in this area.

DETAILED DESCRIPTION:
Nontuberculous mycobacteria are environmental organisms primarily found in soil and water, including locations such as lakes, rivers, agricultural zones, and some industrial sites. Environmental changes facilitate the transport of these organisms to many different settings, including external and internal living spaces. NTM are separate from the Mycobacterium tuberculosis complex (the cause of tuberculosis) and are not the mycobacteria that cause leprosy. With around 200 species, these organisms can be classified into slow growing mycobacteria (SGM ≥ 7 days) or rapid growing mycobacteria (RGM < 7 days), based on their growth rate in solid culture medium. M. avium, M. kansasii, M. xenopi, and M. abscessus are the most common NTM species that can cause pulmonary disease. Unlike M. tuberculosis these mycobacteria are not pathogens, but in the right setting, they can infect humans and produce clinical disease. This is most often seen in people with pre-existing lung damage due to bronchiectasis, chronic obstructive pulmonary disease (COPD), or cystic fibrosis, and NTM infection results in worsening health, and the development of a chronic respiratory illness, NTM-PD.

This study is designed to explore the impact of non-tuberculous mycobacteria-pulmonary disease (NTM-PD) on patients' health, to explore what symptoms are of most concern to people with NTM-PD and to better characterise what non-pharmacological interventions might help this patient group.

The study questions guiding this research are:

1. What are the key clinical differences between people living with NTM pulmonary disease and people with bronchiectasis?
2. What symptoms are of most importance to people with NTM-PD and is this different to people with bronchiectasis?
3. Does the need for non-pharmacological intervention differ for people with NTM-PD compared to other patients with bronchiectasis without NTM-PD? This will be done by comparing the symptoms, investigation results and physiological measurement of people with NTM-PD to a group at risk of NTM-PD but without either NTM infection or disease, namely people with bronchiectasis but no evidence for NTM pulmonary infection. By identifying and analysing any differences between these groups, the study aims to increase the understanding of NTM-PD and so contribute to the development of more effective and evidence-based clinical practice.

This will be accomplished by integrating validated Patient-Reported Outcome Measures (PROMs) with radiological evaluation and respiratory assessments. Additionally, a self-reported questionnaire will be used to rank the most significant symptoms associated with NTM-PD, as well as the daily living activities affected, from the patients' perspective.

The findings could reveal key differences in clinical features and symptoms between these groups, helping to optimise non-pharmacological interventions, improve treatment plans for people with NTM-PD, and highlight areas for future research.

ELIGIBILITY:
Inclusion Criteria:

- Age: 18 years or older, able to provide informed consent.

NTM-PD Group:

* Participants will be adults diagnosed with confirmed NTM-PD based on the British Thoracic Society (BTS) guidelines.
* The participant should not be on any antimicrobial therapy (at least two weeks before participation) and should not have previously received or be currently on antimicrobial therapy for NTM-PD.

  * BTS guidelines:
* Clinical (both required):
* Pulmonary symptoms, nodular or cavitary opacities on chest radiograph, or a high-resolution CT scan that shows multifocal bronchiectasis with multiple small nodules.
* Appropriate exclusion of other diagnoses.
* Microbiological:
* A minimum of two positive expectorated sputum culture results of the same NTM species from samples collected on separate days within 12 months before recruitment.

OR

* Positive culture results from at least one bronchial wash or lavage. OR
* Transbronchial or other lung biopsy with mycobacterial histopathological features (granulomatous inflammation or AFB) and positive culture for NTM or biopsy showing mycobacterial histopathological features (granulomatous inflammation or AFB) and one or more sputum or bronchial washings that are culture-positive for NTM.

Bronchiectasis Group:

* Diagnosed with bronchiectasis, as confirmed in medical records based on clinical assessment, and radiological findings.
* Never had a history of positive culture result for NTM pulmonary infection.
* The latest NTM-negative result must be within the past 12 months from the study's start date or no earlier than 2024.

Exclusion Criteria:

- Age: Under 18 years of age, or unable to provide informed consent.

NTM-PD Group:

* No confirmation of NTM-PD diagnosis.
* Diagnosed with a reinfection of NTM-PD.
* Started antimicrobial therapy for NTM-PD.

Bronchiectasis Group:

* No diagnosis of bronchiectasis or diagnosis of bronchiectasis with NTM-PD.
* Diagnosed with other chronic respiratory diseases considered primary conditions, rather than bronchiectasis.
* Participants with a history of NTM pulmonary infection.
* NTM-negative results obtained before 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Participants diagnosed with NTM-PD.
  * Participants diagnosed with bronchiectasis without NTM pulmonary infection.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | Baseline (during the past week)
  The Quality of Life - Bronchiectasis (QoL-B) questionnaire will be used to assess health-related quality of life of both groups.
  The Qol-B consist of 37 items questionnaire evaluating eight domains (physical function, role function, vitality, emotional function, social functions, treatment burden, health perception, and respiratory symptoms), each scored on a scale from 0 to 100, where higher score indicate better quality of life.

SECONDARY OUTCOMES:
Nutritional Status | Baseline (during the past 3 months)
  Mini Nutritional Assessment (MNA) will be used to assess nutritional status. The MNA consists of 6 items, each score to give a total score range of 0 to 14, where higher scores indicate better nutritional status.
Level of depression | Baseline (during the past 2 weeks)
  The Patient Health Questionnaire-9 (PHQ-9) will be used to screen for the level of depression.
  The PHQ-9 consists of 9 items, each scored from 0 to 3, giving a total score range of 0 to 27, where higher scores indicate higher level of depressive symptoms.
Breathlessness | Baseline (Day of study visit)
  The Modified Medical Research Council Dyspnea Scale (mMRC) will be used to assess the level of breathlessness.
  The mMRC is a 5-point scale ranging from 0 to 4, where higher scores indicate more severe breathlessness.
Lung function test | The most recent test done within the past 2 years.
  Lung function will be assessed using routinely collected spirometry results.
  The following parameters will be collected:
  1. Forced Vital Capacity (FVC): maximum exhaled volume after full inspiration, in litres (L).
  2. Forced Expiratory Volume in one second (FEV₁): volume exhaled in the first second of forced expiration, in litres (L).
  3. FEV₁/FVC ratio: proportion of FVC exhaled in the first second, in percent (%).
  4. Forced Expiratory Flow 25-75% (FEF₂₅-₇₅%): average flow during the middle half of forced expiration, in litres per second (L/sec).
  5. Peak Expiratory Flow Rate (PEFR): maximum flow during forced expiration,in litres per second (L/sec).
  6. Tidal volume (VT): volume inhaled or exhaled during normal breathing, litres (L).
  7. Vital Capacity (VC): maximum exhaled volume after full inspiration, in litres (L).
  Lower results reflect reduced lung function.
Respiratory muscle strength | Baseline (Day of study visit)
  Sniff Nasal Inspiratory Pressure (SNIP) test will be conducted to assess diaphragm and inspiratory muscle strength.
Physical Activity | Baseline (Day of study visit)
  6-minute walk test (6MWT) will be conducted to assess exercise capacity and physical activity.
Body composition | Baseline (Day of study visit)
  Bio-electrical Impedance Analysis (BIA) will be conducted to assess body composition.
  The BIA device will provide the following measures:
  * Fat-free mass (FFM): measured by the device, reported in kilograms (kg).
  * Body fat percentage: calculated by the device as the proportion of fat mass relative to total body weight, reported in percent (%).
  * Fat-free mass index (FFMI): calculated by the device as FFM divided by height squared, reported in kilograms per square metre (kg/m²).
  * Total body water (TBW): estimated by the device from conductivity of body tissues, repoted as volume in litres (L) and as the proportion of total body weight in percent (%).
  Lower FFM, FFMI, or TBW values indicate reduced nutritional or hydration status.
Lung condition | The most recent CT scan done within the past 2 years.
  Radiological scans will be reviewed to assess the extent and pattern of the lung condition.

OTHER OUTCOMES:
Daytime sleepiness | Baseline (during the past week)
  Epworth Sleepiness Scale (ESS) will be used to assess daytime sleepiness and help identify risk for obstructive sleep apnoea (OSA).
  The ESS consists of 8 items, each scored from 0 to 3, giving a total score range of 0 to 24, where higher scores indicate greater daytime sleepiness. A score of 11 or above suggests increased daytime sleepiness.
Obstructive Sleep Apnoea (OSA) | Baseline (during the past week)
  STOP-Bang questionnaire will be used to screen for risk of obstructive sleep apnoea (OSA).
  The acronym STOP-Bang refers to the eight items assessed: Snoring, Tiredness during daytime, Observed apnoea, high blood Pressure, Body mass index, Age, Neck circumference, and Gender.
  The STOP-Bang consists of 8 yes/no items, giving a total score range of 0 to 8, where higher scores indicate a greater risk of OSA.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sulaiman N, Martins B, Moreira-Sousa D, Aguiar A, Hurst JR, Brown J, Duarte R, Lipman M. Optimising non-pharmacological interventions in people with non-tuberculous mycobacterial pulmonary disease: a systematic review. ERJ Open Res. 2025 Dec 22;11(6):00533-2025. doi: 10.1183/23120541.00533-2025. eCollection 2025 Nov. PMID 41438867
- [Background] Ratnatunga CN, Lutzky VP, Kupz A, Doolan DL, Reid DW, Field M, Bell SC, Thomson RM, Miles JJ. The Rise of Non-Tuberculosis Mycobacterial Lung Disease. Front Immunol. 2020 Mar 3;11:303. doi: 10.3389/fimmu.2020.00303. eCollection 2020. PMID 32194556
- [Background] Winthrop KL, Marras TK, Adjemian J, Zhang H, Wang P, Zhang Q. Incidence and Prevalence of Nontuberculous Mycobacterial Lung Disease in a Large U.S. Managed Care Health Plan, 2008-2015. Ann Am Thorac Soc. 2020 Feb;17(2):178-185. doi: 10.1513/AnnalsATS.201804-236OC. PMID 31830805
- [Background] Chalmers JD, Polverino E, Crichton ML, Ringshausen FC, De Soyza A, Vendrell M, Burgel PR, Haworth CS, Loebinger MR, Dimakou K, Murris M, Wilson R, Hill AT, Menendez R, Torres A, Welte T, Blasi F, Altenburg J, Shteinberg M, Boersma W, Elborn JS, Goeminne PC, Aliberti S; EMBARC Registry Investigators. Bronchiectasis in Europe: data on disease characteristics from the European Bronchiectasis registry (EMBARC). Lancet Respir Med. 2023 Jul;11(7):637-649. doi: 10.1016/S2213-2600(23)00093-0. Epub 2023 Apr 24. PMID 37105206
- [Background] Kunst H, Wickremasinghe M, Wells A, Wilson R. Nontuberculous mycobacterial disease and Aspergillus-related lung disease in bronchiectasis. Eur Respir J. 2006 Aug;28(2):352-7. doi: 10.1183/09031936.06.00139005. Epub 2006 Apr 12. PMID 16611651
- [Background] Lipman M, Kunst H, Loebinger MR, Milburn HJ, King M. Non tuberculous mycobacteria pulmonary disease: patients and clinicians working together to improve the evidence base for care. Int J Infect Dis. 2021 Dec;113 Suppl 1:S73-S77. doi: 10.1016/j.ijid.2021.03.064. Epub 2021 Mar 26. PMID 33781905
- [Background] Haworth CS, Banks J, Capstick T, Fisher AJ, Gorsuch T, Laurenson IF, Leitch A, Loebinger MR, Milburn HJ, Nightingale M, Ormerod P, Shingadia D, Smith D, Whitehead N, Wilson R, Floto RA. British Thoracic Society guidelines for the management of non-tuberculous mycobacterial pulmonary disease (NTM-PD). Thorax. 2017 Nov;72(Suppl 2):ii1-ii64. doi: 10.1136/thoraxjnl-2017-210927. No abstract available. PMID 29054853